CLINICAL TRIAL: NCT00448097
Title: A Randomized Study of Cetuximab or Cetuximab Plus Docetaxel Followed by Radical Prostatectomy for Patients With Adenocarcinoma of the Prostate
Brief Title: Efficacy and Safety Study of Cetuximab or Cetuximab Plus Docetaxel to Treat Prostate Cancer Before Prostatectomy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of patient population - slow accrual
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMRI IRB#0206-0027; E-VS-ET-2006 (Other: Principal Investigator)
Record Dates: First submitted 2007-03-14; First posted 2007-03-15 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Prostatic Neoplasms
Keywords: Adenocarcinoma of the Prostate; Prostate cancer; Pre-Prostatectomy; Neoadjuvant
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cetuximab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Data not available PI relocated (Other): No verifiable data available, PI relocated
  Interventions: Drug: cetuximab; Drug: docetaxel

INTERVENTIONS:
Drug: cetuximab — No verifiable data available, PI relocated
  Other Names: Erbitux
Drug: docetaxel — No verifiable data available, PI relocated
  Other Names: Taxotere

SUMMARY:
The purpose of this study is to differentiate between the administrations of Cetuximab alone vs. Cetuximab plus Docetaxel in the treatment of non-metastatic prostate cancer before the surgical removal of the prostate.

DETAILED DESCRIPTION:
With the larger number of men who undergo screening with assays for serum prostate specific antigen, urologists continue to see considerable numbers of patients with locally advanced prostate disease. There is a higher risk of treatment failure in any patient with a tumor that extends through the prostate capsule, more aggressive pathology (Gleason score of 7 or higher), or patients with a PSA of greater than 10 ng/ml. The rationale for adding molecular targeted drugs such as Cetuximab (epithelial growth factor inhibitor), with or without chemotherapy such as Docetaxel, is that such therapy has the potential to demonstrate tumor shrinkage of the prostate and, in addition, micrometastatic cells. Cetuximab alone or Cetuximab plus Docetaxel utilizing the preprostatectomy model, with the adjuvant delivery of Cetuximab for 6 months, will provide data for the following points:

1. demonstration of a PSA response prior to prostatectomy;
2. demonstration whether a change in the natural history, with a delay in the onset of metastatic disease in patients with advanced local prostate cancer, can be achieved;
3. laboratory and tissue correlation to assess changes in proliferative, apoptosis, and pathologic parameters; and
4. metabolic imaging utilizing CT-PET with FDG to assess whether this will be a useful modality in exhibiting a response to therapy, compared with conventional radiographic imaging.

This will provide the basis for future development of neoadjuvant chemotherapy prior to prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of prostatic adenocarcinoma without evidence of regional and/or distant metastasis, clinical stage T1c or T2a with high grade disease (Gleason's 8-10) on initial biopsy, or clinical stage T2b-T2c with Gleason's grade 7 or above with a PSA ≥ 10ng/ml, or clinical stage T3.
* Recent (< 6 weeks prior to study entry) negative bone scan and MRI of abdomen and pelvis.
* Appropriate surgical candidate for radical prostatectomy and a performance status of < 2 (Zubrod scale).
* Patients should have adequate bone marrow function defined as an absolute peripheral granulocyte count > 1,500 and platelet count of > 100,000, adequate hepatic function with a bilirubin < 1.5 mg % and SGPT < 2.5x the upper limits of normal, adequate renal function defined as serum creatinine < 1.5 x ULN.
* Patients must have normal coagulation profile (PT, PTT) and no history of substantial non-iatrogenic bleeding diatheses. Use of anticoagulants is limited to local use only (for control of central line patency).
* Patients must have no history of congestive heart failure or previous MI within the last 12 months.

Exclusion Criteria:

* Previous or current hormonal treatment, chemotherapy, radiation therapy, immunotherapy or other investigational status drug.
* Unable to tolerate transrectal ultrasound.
* Patients who are not appropriate surgical candidates for radical prostatectomy based on the evaluation of co-existent medical diseases and competing causes of death. Patients with uncontrolled cardiac, hepatic, renal or neurologic/psychiatric disorder are not eligible. Patients with uncontrolled and symptomatic orthostatic hypotension or uncontrolled hypertension are not eligible.
* Patients who are HIV positive or have chronic hepatitis B or C infections are not eligible.
* Patients on oral steroid medications are not eligible.
* Patients with significant arteriosclerotic disease, as defined by a previous arterial bypass claudication limiting activity, or a history of cerebrovascular events within the last year (including TIA) are not eligible.
* Prior severe infusion reaction to a monoclonal antibody.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-02; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Pathological response (prostate biopsy vs. prostatectomy specimen pathological evaluation): done pre-treatment vs. after prostatectomy at Week 10 | during study
  No verifiable data available, PI relocated
Clinical response: digital rectal exam pre-treatment and q 6 months after prostatectomy | during study
  No verifiable data available, PI relocated

SECONDARY OUTCOMES:
PSA response: tested q 3 weeks pre-prostatectomy and q 6 months post-prostatectomy | during study
  No verifiable data available, PI relocated
Correlation with MRI and nuclear imaging: scans pre-treatment vs. Week 10 before surgery and yearly when PSA > 0.3 | during study
  No verifiable data available, PI relocated
Correlation with metabolic imaging (PET with FDG): scans pre-treatment vs. Week 10 before surgery | during study
  No verifiable data available, PI relocated
Correlation with serum and plasma for antiangiogenic factors: tested q 3 weeks pre-prostatectomy | during study
  No verifiable data available, PI relocated

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Amato, DO, Principal Investigator — Baylor College of Medicine - Methodist Hospital
Locations (1):
- Baylor College of Medicine - Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prewett M, Rockwell P, Rockwell RF, Giorgio NA, Mendelsohn J, Scher HI, Goldstein NI. The biologic effects of C225, a chimeric monoclonal antibody to the EGFR, on human prostate carcinoma. J Immunother Emphasis Tumor Immunol. 1996 Nov;19(6):419-27. doi: 10.1097/00002371-199611000-00006. PMID 9041461